CLINICAL TRIAL: NCT07215052
Title: Effects of a Suspension Training Warm-up on Cardiopulmonary Exercise Performance in Recreationally Active College-Aged Adults: a Randomized, Counterbalanced Crossover Study
Brief Title: Effects of a Suspension Training Warm-up on Cardiopulmonary Exercise Performance
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tamara Rial-Faigenabum (Other)
Responsible Party: Sponsor-Investigator, Tamara Rial-Faigenabum, Principal Investigator, Coordinator Human Performance Lab and Specialist Professor Monmouth Unversity, Human Performance Lab of Monmouth University
Organization: Human Performance Lab of Monmouth University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SP2553
Record Dates: First submitted 2025-10-08; First posted 2025-10-10 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Exercise Performance
Keywords: cardiorespiratory fitness; exercise physiology

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Walking Warm-up (WW) (Active Comparator): 6 min treadmill walking at comfortable pace, 0% incline.
  Interventions: Other: Walking Warm-up
- Suspension Warm-up (SW) (Experimental): 6 min dynamic TRX warm-up (reverse lunges, squats, jump squats, rows, push-ups).
  Interventions: Other: Suspension Training Warm-up

INTERVENTIONS:
Other: Walking Warm-up — 6 minutes treadmill walking at comfortable self-selected pace, 0% incline.
  Arms: Arm 1: Walking Warm-up (WW)
Other: Suspension Training Warm-up — 6 minutes TRX suspension warm-up (reverse lunges 45s, squats 60s, jump squats 45s, rows 30s, push-ups 30s, with 30s rests).
  Arms: Suspension Warm-up (SW)

SUMMARY:
this study will compare two warm-up methods before cardiopulmonary exercise testing (CPET) in recreationally active young adults. Participants will complete treadmill walking or TRX suspension warm-up, followed by a treadmill exercise test to exhaustion. The investigators to determine whether suspension warm-up produces similar peak oxygen uptake (VO2max) and cardiopulmonary responses as treadmill walking.

DETAILED DESCRIPTION:
CPET is the gold standard for assessing aerobic fitness. Warm-up procedures may influence outcomes. Traditional CPET warm-up uses walking or cycling, but suspension training provides a dynamic, full-body option. This randomized, counterbalanced crossover study will compare VO₂max and secondary outcomes (time to exhaustion, HRmax, RER, VE, BP, VT) after treadmill vs suspension training warm-up. The primary analysis is a non-inferiority test with a 5% margin for VO₂max.

ELIGIBILITY:
Inclusion Criteria:

Aged 19 to 25 years

Engages in ≥5 hours per week of moderate-to-vigorous physical activity (classified as "high activity" based on the International Physical Activity Questionnaire [ICIQ])

Able to pass the Physical Activity Readiness Questionnaire (PAR-Q+) screening

Exclusion Criteria:

Participates in <5 hours per week of moderate-to-vigorous physical activity

Contraindications to maximal cardiopulmonary exercise testing or suspension training

Presence of any medical condition that may interfere with safe test participation or data interpretation

-

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
VO₂peak (mL·kg-¹·min-¹) | Immediately following each warm-up condition during two laboratory visits, separated by at least 48 hours
  VO₂peak measured during cardiopulmonary exercise testing (CPET) following each warm-up condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Monmouth University Graduate Center Room 222, West Long Branch, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be made publicly available because this is a small, single-site academic study conducted for exploratory purposes, and data sharing is not required by the sponsor or funding agency. Summary results will be posted on ClinicalTrials.gov and may be included in peer-reviewed publications.